CLINICAL TRIAL: NCT03688789
Title: Prevalence of Adrenal Insufficiency Post-chemotherapy Adrenocorticotropia in Adult Hematology
Brief Title: Hématologie Adulte Prevalence of Adrenal Insufficiency Post-chemotherapy Adrenocorticotropia in Adult Hematology
Acronym: HemaSur
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator leaving the hospital
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC17_8996_HemaSur
Record Dates: First submitted 2018-09-20; First posted 2018-09-28 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Haematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydrocortisone supplementation (Experimental)
  Interventions: Other: Hydrocortisone supplementation

INTERVENTIONS:
Other: Hydrocortisone supplementation — * Cortisol at T0 and T30 mins less than 550 nmol / L after ACTH 250 μG achieved during the last chemotherapy session
  * Hydrocortisone supplementation in patients with biological adrenal insufficiency
  * scale of quality of life estimated by EORTC QLQ-C30

SUMMARY:
A recent meta-analysis involving 3753 patients treated with corticosteroids notes that the population with the highest prevalence of biological IS (68%) is onco-hematology. However, it is also the least studied population with no recent and significant prevalence study. A recent multicenter study including patients followed up oncology who received dexamethasone for antiemetic purposes at cumulative doses well below the doses used in Hematology, objective a prevalence of biological IS estimated at 16% at 3 months from the start of chemotherapy. The introduction of a substitution had led to an objective improvement in the quality of life estimated by EORTC QLQ-C30.

DETAILED DESCRIPTION:
A recent meta-analysis involving 3753 patients treated with corticosteroids notes that the population with the highest prevalence of biological IS (68%) is onco-hematology. However, it is also the least studied population with no recent and significant prevalence study. A recent multicenter study including patients followed up oncology who received dexamethasone for antiemetic purposes at cumulative doses well below the doses used in Hematology, objective a prevalence of biological IS estimated at 16% at 3 months from the start of chemotherapy. The introduction of a substitution had led to an objective improvement in the quality of life estimated by EORTC QLQ-C30.

Expected results are prevalence rate of biological adrenal insufficiency between 15 and 20% with improvement of the quality of life in the 2 months post-chemotherapy by Hydrocortisone supplementation

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Patient naive to any chemotherapy treatment, re-ceiving a 1st chemotherapy line of RCHOP, RCOP, VTD, VD or MPT type from the Adult Hematology Department
* PS according to WHO = 0,1 and 2

Exclusion Criteria:

* Adrenal pathology, hypothalamus or pre-existing pituitary gland (including metastatic lesions)
* Long-term treatment with corticosteroids or in the previous 6 months
* Refusal or absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Cortisol at T0 and T30 mins less than 550 nmol / L after ACTH 250 μG achieved during the last chemotherapy session | 30 min
  Cortisol at T0 and T30mins less than 550 nmol / L after ACTH 250 μG achieved during the last chemotherapy session

SECONDARY OUTCOMES:
cumulative doses of corticosteroids in prednisone equivalent as well as duration of exposure | 6 months
  cumulative doses of corticosteroids in prednisone equivalent as well as duration of exposure
potential drug interactions (including CYP450 inducer) | 6 months
  potential drug interactions (including CYP450 inducer)
Evaluation of the effect on quality of life of Hydrocortisone supplementation in patients with biological IS in the wake of EORTC QLQ-C30 type self-administered chemotherapy at D0 and D30 | 30 days
  Evaluation of the effect on quality of life of Hydrocortisone supplementation in patients with biological IS in the wake of EORTC QLQ-C30 type self-administered chemotherapy at D0 and D30

CONTACTS AND LOCATIONS:
Overall Officials: Brieuc Cherel, MD, Principal Investigator — Rennes University Hospital